CLINICAL TRIAL: NCT03369171
Title: Wearable Biosensor to Track and Quantify Limb Dysfunction in Multiple Sclerosis Patients
Acronym: MYO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RC16_0391
Record Dates: First submitted 2017-10-31; First posted 2017-12-11 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with MYO armband (Experimental)
  Interventions: Device: Myo Armband (MYO,Thalamic Labs Inc, Kitchener, ON, Canada)

INTERVENTIONS:
Device: Myo Armband (MYO,Thalamic Labs Inc, Kitchener, ON, Canada) — MYO armband is a commercialized, gesture control device containing "Height Medical Grade Stainless Steel EMG sensors", and an inertial measurement unit (IMU) consisting of a three-axis gyroscope and a, three-axis accelerometer, three-axis magnetometer. MY0 motion data (EMG and IMU) will be recorded during standard motor/neurological evaluation.
  The clinical assessment will include standard motor neurological evaluation : EDSS and FS, walking status, foot tapping test, Heel-knee test, finger tapping test, Finger to nose test, Romberg test, timed 25 foot walk test, nine holes peg test. This clinical assessment will be done at the inclusion visit (V1) and at the follow-up visit at one year (V2).
  Other Names: MYO, Gesture control armband

SUMMARY:
Multiple sclerosis (MS) is a leading cause of neurological injury in young adults. Capturing the extent of multiple domains of MS-related disability is critical for effective clinical care and the development of new paradigms for patient-focused therapeutic approaches. To date outcomes research in MS has centered on clinical exams, which may be insensitive over the short term (the 1-2 years of early stage clinical trials) and only capture a single snapshot of the patient's performance.

With the mass production of sensors in the gaming and computer control industry, there is an opportunity to transform the traditional neurological exam with biosensors already in use outside the realm of health applications. The investigators herein propose to use a commercialized wearable electroMYOgraphy sensor (MYO,Thalamic Labs Inc, Kitchener, ON, Canada) for detection of upper and lower limb dysfunction in MS patients. The investigators will determine if the device can differentiate the diseased states, refine signal processing algorithms to create reliable outcomes using this device in MS patients, and determine if these outcomes are strongly associated with patients and physicians reported ambulatory and dexterity metrics. The investigators hypothesize that this digital technology may be introduced in the standard neurological exam technique in a non-disruptive manner and more accurately and potentially remotely detect both physician-reported and patient-reported disability.

In the scope of this study, the investigators will also develop signal processing methodology to comprehensively track ambulation features.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a leading cause of neurological injury in young adults. Capturing the extent of multiple domains of MS-related disability is critical for effective clinical care and the development of new paradigms for patient-focused therapeutic approaches. To date outcomes research in MS has centered on clinical exams, which may be insensitive over the short term (the 1-2 years of early stage clinical trials) and only capture a single snapshot of the patient's performance.

With the mass production of sensors in the gaming and computer control industry, there is an opportunity to transform the traditional neurological exam with biosensors already in use outside the realm of health applications. The investigators herein propose to use a commercialized wearable electroMYOgraphy sensor (MYO,Thalamic Labs Inc, Kitchener, ON, Canada) for detection of upper and lower limb dysfunction in MS patients. The investigators will determine if the device can differentiate the diseased states, refine signal processing algorithms to create reliable outcomes using this device in MS patients, and determine if these outcomes are strongly associated with patients and physicians reported ambulatory and dexterity metrics. The investigators hypothesize that this digital technology may be introduced in the standard neurological exam technique in a non-disruptive manner and more accurately and potentially remotely detect both physician-reported and patient-reported disability.

In the scope of this study, the investigators will also develop signal processing methodology to comprehensively track ambulation features.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 to 64 years inclusive (Patients over 64 years will not be enrolled to avoid possible effect of aging on the voluntary movement assessed);
* Confirmed diagnosis of MS according to the revised McDonald criteria (including primary progressive, secondary progressive and relapsing-remitting MS) with brain lesions consistent with MS if data available;
* No history of relapse in the previous 5 weeks.
* Must be able or think they are able to attempt both finger and foot tapping tests, F2NT, 9HPT and be ambulatory with or without assistance.

Exclusion Criteria:

* Pregnant women
* Minors
* Adults under guardianship
* Adults over 64 years

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2018-01-23 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Discrimination of walking disorder status | Day 0
  Normal or Abnormal walking status of MS patients will be determined at baseline based on clinical judgement and compared to EMG data from calf muscle of the more affected limb combined with Inertial Motion Unit (IMU).

SECONDARY OUTCOMES:
Foot tapping test | day 0
  [Foot tapping test is used to assess rapid alternating movement of the lower extremity and coordination]. Each lower extremity is assessed separately (by neurologist) while MYO is placed over calf muscle. Foot tapping test result based on clinical judgment is compared to MYO motion data.
Finger tapping test | day 0
  [Finger tapping test is used to assess rapid alternating movement of the upper extremity and coordination]. Each extremity is assessed separately (by neurologist) while MYO is placed over forearm muscle. Finger tapping test result based on clinical judgment is compared to MYO motion data.
Heel-knee test | day 0
  : [Heel knee test is used to assess coordination of lower extremities and to detect cerebellum dysfunction]. Each extremity is tested separately (by neurologist) while MYO is placed over calf muscle. Heel-knee test result based on clinical judgment is compared to MYO motion data
Romberg test | day 0
  The Romberg test is used to assess balance. The test is performed while the patient is wearing MYO on the calf of the most affected leg
Finger to nose test | day 0
  [Finger to nose test is used to assess coordination of upper extremity movement]. Each extremity is assessed separately (by neurologist) while MYO is placed over forearm muscle. Finger to nose test result based on clinical judgment is compared to MYO motion data
Timed 25 foot walk test result | day 0
  Timed 25 foot walk (T25FW) is used to measure walking function based on time. T25FW is a quantitative mobility and leg function performance test. Patient is asked to walk 25 feet with MYO device placed over calf muscle of the most affected leg
Nine holes peg test | day 0
  The nine holes peg test (9-HPT) is used to measure fine manual dexterity. 9-HPT measures the time it takes to place 9 pegs into 9 holes and then remove the pegs. Each side is tested separately with MYO placed over forearm muscle. Ability of MYO sensor to detect upper dysfunction is evaluated.
Expanded disability status scores (EDSS) | Day 0 and at one year
  EDSS is a 20-step ordinal scale of disease severity ranging from to 10 in 0.5 increments (when reaching EDSS 1), with higher scores indicating more disability. Scoring is based on assessment by a neurologist of clinical deficit (rate from 0 to 5 or 6) in 8 functional systems (FS) combined with ambulation ability/mobility
Patient-reported disability using self-report questionnaire | Day 0 and at one year
  The questionnaire comprises 17 questions related to MS. To study the relationship between MYO motion data and patient-perceived disability
Twelve items Multiple Sclerosis Walking Scale Assessment (MSWS-12) scale | Day 0 and at one year
  : MSWS-12 is a 12-item patient rate measure of the impact of MS on the individual's walking ability during the past 2 weeks. Each item is rate from 1 (no difficulty) to 5 (extreme difficulty) then summed (ranging from 12 to 60, with higher score reflecting a greater impact of MS on walking). To study the relationship between MYO motion data and patient-perceived mobility.
12-item version of World Health Organization Disability Assessment Schedule (WHODAS 2.0) | Day 0 and at one year
  The short version of WHODAS 2.0 comprises 12 questions related to difficulties experienced in six domains (mobility, self-care, life activities, understanding and communicating interpersonal interactions, and participation in society) during the previous 30 days. Each item is rated from 1 (no problem) to 5(extreme). The scores from each item are summed to generate a total score ranging from 12 to 60, with higher score reflecting higher levels of disability. To study the relationship between MYO motion data and quality of life (related to disability)
Disability as measured with EDSS score | Day 0 and at one year
  To study the relationship between MYO motion data and physician-scored rated disability
Disability as measured with Functional systems score (FS) | Day 0 and at one year
  To study the relationship between MYO motion data and physician-scored rated disability
Dysfunction assessed by walking disorder status | Day 0 and at one year
  Dysfunction assessed by clinical exam of walking disorder status is compared to MYO motion data.
Dysfunction assessed by foot tapping test | Day 0 and at one year
  Dysfunction assessed by clinical exam of foot tapping test is compared to MYO motion data.
Dysfunction assessed by finger tapping test | Day 0 and at one year
  Dysfunction assessed by clinical exam of finger tapping test is compared to MYO motion data.
Dysfunction assessed by heel-knee test | Day 0 and at one year
  Dysfunction assessed by clinical exam of heel-knee test is compared to MYO motion data.
Dysfunction assessed by Romberg test | Day 0 and at one year
  Dysfunction assessed by clinical exam of Romberg test is compared to MYO motion data.
Dysfunction assessed by finger to nose test | Day 0 and at one year
  Dysfunction assessed by clinical exam of finger to nose test is compared to MYO motion data.
Dysfunction assessed by timed 25 foot walk test result | Day 0 and at one year
  Dysfunction assessed by clinical exam of timed 25 foot walk test is compared to MYO motion data.
Dysfunction assessed by nine holes peg test | Day 0 and at one year
  Dysfunction assessed by clinical exam of nine holes peg test is compared to MYO motion data.

CONTACTS AND LOCATIONS:
Overall Officials: David Laplaud, PU-PH, Principal Investigator — Nantes University Hospital
Locations (1):
- CHU de Nantes, Nantes, France